CLINICAL TRIAL: NCT07324395
Title: Delayed Onset Muscle Soreness in the Gastrocnemius Alters Biomechanical, Viscoelastic Properties, and Trunk Endurance in the Posterior Chain Muscles
Brief Title: Posterior Chain Responses to Gastrocnemius DOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ebru Aloğlu Çiftçi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ebru Aloğlu Çiftçi, PhD student, Istinye University
Organization: Istinye University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GDYY01
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Delayed Onset Muscle Soreness (DOMS); Healthy
Keywords: Delayed onset muscle soreness; posterior chain muscles; Trunk Endurance; muscle stiffness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOMS Induction Arm (Experimental): Participants in this arm will complete a standardized exercise protocol designed to induce delayed onset muscle soreness (DOMS) in the gastrocnemius muscle. All assessments will be performed at baseline, immediately after the DOMS protocol, and at 24, 48, and 72 hours.
  Interventions: Other: Gastrocnemius DOMS Induction Protocol

INTERVENTIONS:
Other: Gastrocnemius DOMS Induction Protocol — Participants will complete an eccentric exercise protocol to safely induce delayed onset muscle soreness (DOMS) in the gastrocnemius muscle. The protocol includes:
  Exercise performed bilaterally, starting with the dominant leg Three sets of eccentric heel-lowering movements A 5-minute rest period between sets Participants place the foot on a step and lower the heel for 3 seconds using eccentric contraction The heel is lowered until no further downward motion is possible The opposite leg is used only to lift the body back to the starting position in 1 second A metronome set to 60 beats per minute is used to control movement speed Each set ends when the participant can no longer maintain the required tempo Participants are instructed to avoid physical activity and not take any pain-relieving medication during the 72-hour follow-up period.
  Intervention Model Description: All participants receive the same DOMS induction protocol.

SUMMARY:
The goal of this clinical trial is to learn how delayed onset muscle soreness (DOMS) in the calf muscle (gastrocnemius) affects the muscles of the posterior chain and physical performance in healthy young adults. The main questions the study aims to answer are:

Does DOMS in the calf muscle change the biomechanical properties (tone, stiffness, elasticity) of other muscles in the posterior chain?

Does DOMS lower trunk endurance, muscle strength, balance, or jump performance?

Participants will:

Take part in a gastrocnemius exercise protocol designed to safely create DOMS

Complete repeated assessments at baseline, immediately after exercise, and at 24, 48, and 72 hours

Have their muscle properties measured with a handheld device

Complete trunk endurance tests, muscle strength tests, balance tests, and a vertical jump test

Provide a blood sample to measure creatine kinase (a marker of muscle damage)

This research may help clinicians better understand how soreness in one muscle can influence the whole posterior chain and may guide safer training and recovery strategies.

DETAILED DESCRIPTION:
This prospective repeated-measures clinical trial includes healthy adults aged 18-25 years. DOMS will be induced using a standardized exercise protocol targeting the gastrocnemius muscle. Outcome measures will be collected at five time points: baseline, immediately after the DOMS-inducing exercise, and 24, 48, and 72 hours post-exercise.

Primary outcomes include muscle biomechanical properties such as muscle tone, stiffness, elasticity, relaxation, and creep, measured using a digital myotonometer. Trunk endurance is also assessed as a primary outcome because of the posterior chain's role in load transfer and stabilization.

Secondary outcomes include:

Muscle strength

Dynamic balance performance

Vertical jump height

Pain pressure threshold

Serum creatine kinase levels to confirm muscle damage

To reduce assessment bias, each assessor is responsible for only one measurement type and is blinded to the DOMS-induction procedure. All assessments occur at the same time points for all participants.

The study aims to provide new information about how localized muscle soreness affects chain-related muscle behavior and functional performance. Findings may contribute to improved injury-prevention, training, and rehabilitation strategies, especially for populations exposed to high mechanical load.

ELIGIBILITY:
Inclusion Criteria:

* The study included 14 volunteers aged 18-25 with a resting heart rate between 50 and 90 beats per minute who were right-handed.

Exclusion Criteria:

* Individuals who had undergone lower extremity injury or surgery in the past six months were excluded from the study. Those with chronic lower extremity pain or systemic or neurological diseases were also excluded. Participants with vision or hearing problems that could affect balance were excluded. Individuals who regularly used medication, smoked, consumed alcohol, or used other harmful substances were also excluded. Participants who regularly used caffeine or vitamin C supplements or who had an exercise habit were also excluded from the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Muscle Biomechanical Properties (Muscle Tone) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Muscle tone (F) will be assessed using the MyotonPRO device. Measurements will be recorded in Hertz (Hz). Measurements will be taken three times for each muscle segment, and the average value will be calculated.
  Standardized anatomical landmarks were used for each muscle:
  Gastrocnemius: measured at the thickest part of the medial head, approximately 10 cm below the popliteal crease. The location was confirmed with a tape measure to account for individual differences. Hamstrings: measured with the participant in a prone position, at the midpoint between the ischial tuberosity and the fibular head. Gluteus maximus: measured at the thickest portion of the muscle identified by palpation while the participant was prone. Erector spinae: measured 2.5 cm lateral to the L5 spinous process in the prone position. Measurement points were marked on the skin to en
Muscle Biomechanical Properties (Muscle Stiffness) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Muscle stiffness (S) will be assessed using the MyotonPRO device. Results will be reported in Newtons per meter (N/m).
  Measurements will be taken three times for each muscle segment, and the average value will be calculated. Standardized anatomical landmarks were used for each muscle: Gastrocnemius: measured at the thickest part of the medial head, approximately 10 cm below the popliteal crease. The location was confirmed with a tape measure to account for individual differences. Hamstrings: measured with the participant in a prone position, at the midpoint between the ischial tuberosity and the fibular head. Gluteus maximus: measured at the thickest portion of the muscle identified by palpation while the participant was prone. Erector spinae: measured 2.5 cm lateral to the L5 spinous process in the prone position. Measurement points were marked on the skin to en
Muscle Biomechanical Properties (Muscle Elasticity) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Muscle elasticity will be characterized by the logarithmic decrement (D) measured using the MyotonPRO device. This is a unitless (relative) value representing the ability of the muscle to restore its shape after deformation. Measurements will be taken three times for each muscle segment, and the average value will be calculated. Standardized anatomical landmarks were used for each muscle: Gastrocnemius: measured at the thickest part of the medial head, approximately 10 cm below the popliteal crease. The location was confirmed with a tape measure to account for individual differences. Hamstrings: measured with the participant in a prone position, at the midpoint between the ischial tuberosity and the fibular head. Gluteus maximus: measured at the thickest portion of the muscle identified by palpation while the participant was prone. Erector spinae: measured 2.5 cm lateral to the L5 spinous process in the prone position. Measurement points were marked on the skin to en
Muscle Biomechanical Properties (Muscle Relaxation Time) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Mechanical stress relaxation time (R) will be measured using the MyotonPRO to assess the time the muscle takes to return to rest following deformation. Results will be reported in milliseconds (ms).
  Measurements will be taken three times for each muscle segment, and the average value will be calculated. Standardized anatomical landmarks were used for each muscle: Gastrocnemius: measured at the thickest part of the medial head, approximately 10 cm below the popliteal crease. The location was confirmed with a tape measure to account for individual differences. Hamstrings: measured with the participant in a prone position, at the midpoint between the ischial tuberosity and the fibular head. Gluteus maximus: measured at the thickest portion of the muscle identified by palpation while the participant was prone. Erector spinae: measured 2.5 cm lateral to the L5 spinous process in the prone position. Measurement points were marked on the skin to en
Muscle Biomechanical Properties (Muscle Creep) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Muscle creep will be assessed as the ratio of relaxation and deformation time (Creep (C)) using the MyotonPRO device. This parameter is a relative unit and indicates viscoelastic behavior of the muscle.
  Measurements will be taken three times for each muscle segment, and the average value will be calculated. Standardized anatomical landmarks were used for each muscle: Gastrocnemius: measured at the thickest part of the medial head, approximately 10 cm below the popliteal crease. The location was confirmed with a tape measure to account for individual differences. Hamstrings: measured with the participant in a prone position, at the midpoint between the ischial tuberosity and the fibular head. Gluteus maximus: measured at the thickest portion of the muscle identified by palpation while the participant was prone. Erector spinae: measured 2.5 cm lateral to the L5 spinous process in the prone position. Measurement points were marked on the skin to en
Trunk Endurance Assessment (Sorenson Test) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Sorenson Test: Participants lay prone with their pelvis at the table edge and ankles secured. They held their upper body in a horizontal position, and the time they could maintain the position was recorded. The test ended when the participant could no longer keep the trunk horizontal.
Trunk Endurance Assessment (Sit-up Test) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Sit-up Test: Participants sat with knees flexed at 90° and their upper body positioned at a 60° angle. Arms were crossed over the chest. Time was recorded until the participant's upper body dropped below the 60° angle.
Trunk endurance assessment (Side Bridge Test-Right and Left) | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Participants lay on their side and lifted their hips to form a straight line with the torso. The duration they could maintain this position was recorded. The test was performed on both sides.

SECONDARY OUTCOMES:
Muscle Strength | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Muscle strength of the gastrocnemius, hamstrings, and gluteus maximus was measured using a Lafayette hand-held dynamometer with the "make test" method. The results measured with the dynamometer were recorded in Newtons. Participants pushed against the fixed device with maximal effort for 3-5 seconds in standardized positions:
  Gastrocnemius: foot pushing against the wall in a reverse sit-up position.
  Hamstrings: prone position with the knee at 30° flexion; force applied toward knee flexion.
  Gluteus maximus: prone with knee at 90° flexion; force applied during hip extension.
Dynamic balance performance | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Dynamic balance was assessed using the Y-Balance Test. Participants stood barefoot on the central platform and reached in the anterior, posteromedial, and posterolateral directions while keeping their hands on their hips. Each direction included four practice trials and three test trials for each leg. Reach distances were recorded in centimeters and normalized to leg length. A composite score was calculated using the three reach directions. Leg dominance was determined by asking which leg the participant would use to kick a ball.
Vertical jump test | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  To assess participants' functional performance, a vertical jump test was administered. During the test, participants were asked to jump as high as possible with both feet in front of a platform fixed to the wall. First, the participant's normal arm length was determined by touching the highest point they could reach. Then, participants performed two trials to achieve the highest jump distance, and the best value was recorded. The difference between the jump distance and the normal arm length, calculated in centimeters, was used as a performance measure.

OTHER OUTCOMES:
Creatine Kinase | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  Creatine kinase (CK) levels were measured to confirm muscle damage. Blood samples were collected into heparin tubes and then centrifuged to separate the serum. Serum samples were stored at -80°C until analysis. CK levels were measured using a standard ELISA kit. During the test, serum samples and standards were placed into antibody-coated wells, followed by incubation with biotin and Streptavidin-HRP to form an immune complex. After washing, color-developing solutions were added, and the final color change was measured at 450 nm using a microplate reader. Higher CK values indicate greater muscle damage.
Pain pressure threshold | Baseline, 24 hours post-DOMS, 48 hours post-DOMS, and 72 hours post-DOMS
  The pain pressure threshold (PPT) was assessed using a dolorimeter device. The dolorimeter (Baseline Push-Pull Force Gauge, New York, USA) was applied vertically to the medial and lateral gastrocnemius muscles, increasing by 1 kg/cm² every three seconds until the participant felt pain. This procedure was repeated three times. A minimum of 20 seconds was allowed between measurements, and the average of the measurements was taken. The validity and reliability of the method have been demonstrated in the literature, with a Cronbach's alpha value of 0.84 reported, indicating internal consistency.
Physical Activity Level (IPAQ-Short Form) | Baseline only (assessed once before the DOMS protocol)
  Physical activity levels were assessed at baseline using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The questionnaire consists of 7 items asking participants about the total time spent in light, moderate, and vigorous physical activity during the previous 7 days. Activity scores were calculated by multiplying the time reported for each activity level by its corresponding metabolic equivalent (MET value: 3.3 for light, 4.0 for moderate, and 8.0 for vigorous activity). Total physical activity was recorded as MET-minutes per week. This measure was used as a sociodemographic characteristic and was not reassessed during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Topkapi Campus, Maltepe, Teyyareci Sami St. No:3,, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the ethics approval for this study does not allow external sharing of participant data, even in de-identified form.

REFERENCES:
- [Background] Baird MF, Graham SM, Baker JS, Bickerstaff GF. Creatine-kinase- and exercise-related muscle damage implications for muscle performance and recovery. J Nutr Metab. 2012;2012:960363. doi: 10.1155/2012/960363. Epub 2012 Jan 11. PMID 22288008